CLINICAL TRIAL: NCT02273102
Title: A Phase 1 Dose Escalation Study of Tranylcypromine (TCP) in Combination With ATRA (Tretinoin) for Adult Patients With Relapsed/Refractory Acute Myelogenous Leukemia (AML) and Myelodysplastic Syndromes (MDS)
Brief Title: Study of TCP-ATRA for Adult Patients With AML and MDS
Acronym: TCP-ATRA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Women's Cancer Association (Unknown); Gabrielle's Angel Foundation (Other)
Responsible Party: Principal Investigator, Justin Watts, MD, Assistant Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140328
Record Dates: First submitted 2014-10-20; First posted 2014-10-23 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndromes; Leukemia
Keywords: Acute Myelogenous Leukemia; AML; Myelodysplastic Syndromes; MDS; Tranylcypromine; TCP; ATRA; Tretinoin
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Tranylcypromine; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- TCP Dose Level 1 (Experimental): 20mg of Tranylcypromine (TCP) to be administered orally twice a day (12 hours apart) for up to 16 cycles of 21 days each. 45 mg/m2 of Tretinoin (ATRA) to be administered orally twice a day (12 hours apart) beginning on day 4 of each 21 day cycle, for up to 16 cycles.
  Interventions: Drug: Tranylcypromine; Drug: Tretinoin
- TCP Dose Level 2 (Experimental): 40mg of Tranylcypromine (TCP) to be administered orally twice a day (12 hours apart) for up to 16 cycles of 21 days each. 45 mg/m2 of Tretinoin (ATRA) to be administered orally twice a day (12 hours apart) beginning on day 4 of each 21 day cycle, for up to 16 cycles.
  Interventions: Drug: Tranylcypromine; Drug: Tretinoin
- TCP Dose Level 3 (Experimental): 60mg of Tranylcypromine (TCP) to be administered orally twice a day (12 hours apart) for up to 16 cycles of 21 days each. 45 mg/m2 of Tretinoin (ATRA) to be administered orally twice a day (12 hours apart) beginning on day 4 of each 21 day cycle, for up to 16 cycles.
  Interventions: Drug: Tranylcypromine; Drug: Tretinoin

INTERVENTIONS:
Drug: Tranylcypromine — Tranylcypromine (TCP) to be administered orally twice a day (12 hours apart) for up to 16 cycles of 21 days each.
  Other Names: TCP
Drug: Tretinoin — 45 mg/m2 of ATRA to be administered orally twice a day (12 hours apart), beginning on day 4 for up to 16 cycles of 21 days each.
  Other Names: ATRA

SUMMARY:
Acute Myeloid Leukemia (AML) is a diverse disease that is fatal in the majority of patients. Acute promyelocytic leukemia (APL) however, a subtype of AML accounting for 5% of all cases, is very curable. APL cells are highly sensitive to the retinoid all-trans-retinoic acid (ATRA), which effectively differentiates the leukemic clone. Over 80% of APL patients can be cured with ATRA based therapies. For patients with non-APL AML, ATRA has little effect. Consequently, 85% of these patients will succumb to their disease despite conventional approaches. Little is known about mechanisms of resistance to ATRA in non-APL AML. This knowledge gap limits the use of ATRA in a disease that already has few effective therapies. The investigators' preliminary data suggest that non-APL AML cells can be re-sensitized to ATRA when combined with lysine-specific demethylase 1 (LSD 1) inhibitors. The investigators' publication in Nature Medicine showed that LSD1 inhibition with tranylcypromine (TCP), unlocked the ATRA-driven therapeutic response in non-APL AML. Notably, treatment with ATRA and TCP markedly diminished the engraftment of primary human AML cells in murine models, indicating that the combination may target leukemia-initiating cells (LIC). The investigators' data identify LSD1 as a therapeutic target and strongly suggest that it may contribute to ATRA resistance in non-APL AML. The investigators' central hypothesis is that ATRA combined with TCP will be safe and effective in a clinical population, and that this approach will suppress LICs and restore myeloid differentiation programs in patients with non-APL AML. Testing this hypothesis with the phase I clinical trial outlined in this protocol, will establish a new treatment paradigm in AML and extend the important anti-cancer effects of ATRA to all AML subtypes.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of one of the following:

   * Relapsed/refractory Acute Myelogenous Leukemia (AML) as defined by the World Health Organization (WHO) criteria [therapy-related AML and/or secondary AML from an antecedent hematologic disorder not excluded].
   * Relapsed/refractory Myelodysplasic Syndrome (MDS) as defined by the World Health Organization (WHO) criteria.
2. Adult patients 18 years of age or older.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
4. Adequate organ function as defined as:

   * Total bilirubin ≤ 1.5 x upper limited of normal (ULN)
   * ALT and AST must be ≤ 3 × ULN
   * Creatinine ≤ 1.5 x ULN or calculated creatinine clearance > 50ml/min or
   * PT and aPTT ≤ 1.5 × ULN

     * Patients with total bilirubin, Alanine transaminase (ALT), Aspartate transaminase (AST), Creatinine, prothrombin time (PT), and activated partial thromboplastin time (aPTT) levels outside the permitted range are eligible if, in the judgment of the Principal Investigator, the levels are related to the patient's AML or MDS.
5. Suitable venous access to allow for all study related blood sampling (safety and research).
6. Estimated life expectancy, in the judgment of the Investigator, which will permit receipt of at least 6 weeks of treatment.
7. Able to understand and willing to signed the written informed consent and HIPAA document/s.

Exclusion Criteria:

1. Therapy with moderate or strong CYP3A4 inhibitors or CYP3A4 inducers within 14 days prior to Cycle1 Day1.
2. Therapy with Monoamine Oxidase Inhibitors (MAOIs), dibenzazepine derivatives, sympathomimetics, or Selective Serotonin Reuptake Inhibitors (SSRIs) within 14 days prior to Cycle1 Day1. (Patients actively receiving a safe substitute in the judgment of the Principal Investigator are eligible and may continue to receive the safe substitute during protocol treatment)
3. Therapy with any investigational products, antineoplastic therapy, or radiotherapy within 14 days prior to Cycle1 Day1. Patients actively receiving hydroxyurea are eligible and may continue to receive hydroxyurea during protocol treatment.
4. Candidates for standard and/or potentially curative treatments. (Candidate defined as a patient that is both eligible and willing)
5. Major surgery within 28 days prior to Cycle1 Day1.
6. Grade 2 or higher diarrhea as defined by NCI CTCAE Version 4.03 despite optimal antidiarrheal supportive care within 7 days prior to Cycle1, Day1.
7. Myocardial infarction within 6 months (24 weeks) prior to Cycle1, Day1.
8. Class III or IV heart failure as defined by the New York Heart Association (NYHA), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. (Any ECG abnormality at screening has to be documented by the investigator as not medically relevant and confirmed by the Principal Investigator)
9. Active and uncontrolled infection.
10. Known human immunodeficiency virus (HIV) positive.
11. Known hepatitis B surface antigen-positive.
12. Known or suspected active hepatitis C infections (Patients who are hepatitis C surface antigen-positive are eligible).
13. Female patients who are pregnant women or breast feeding. Confirmation that the patient is not pregnant will require a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women.
14. Females of child bearing potential who refused to either practice 2 effective methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing the informed consent through 30 days after the last dose of study drug.
15. Males of child bearing potential who refuse to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug (includes males surgically sterilized - i.e. status post vasectomy).
16. Serious medical or psychiatric illness/condition likely in the judgment of the Investigator to interfere with compliance to protocol treatment/research.
17. Known history of allergic reaction to TCP or ATRA.
18. Symptomatic central nervous system (CNS) involvement.
19. A concurrent second active and non-stable malignancy (Patients with a concurrent second active but stable malignancy are eligible).
20. Patients with proliferative AML will be excluded defined by a white blood cell count (WBC) > 5 x ULN UNLESS, the white count has been suppressed to < 5 x ULN with hydroxurea and has remained below this level for at least 2 weeks prior to enrollment on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of Toxicity in Study Participants Receiving TCP/ATRA Combination Therapy | 24 months
  The safety and tolerability of TCP/ATRA combination therapy in patients with Acute Myelogenous Leukemia (AML) and Myelodysplastic Syndromes (MDS). This will be measured by the rate of adverse events, serious adverse events and other toxicities in study participants receiving protocol therapy.

SECONDARY OUTCOMES:
Rate of Preliminary Efficacy of TCP/ATRA Combination Therapy | 24 months
  Best response to TCP/ATRA combination therapy will be determined using serial blood and bone marrow sampling throughout the course of treatment. Responses will be documented according to revised/modified International Working Group (IWG) Response Criteria - Cheson et al. 2003 for AML and Cheson et al. 2006 for MDS. Morphologic complete remission (CR), cytogenetic CR, and molecular CR will be assessed by blood counts and simultaneous examination of the bone marrow fpr percentage of bone marrow blasts, as well as cytogenetics and molecular studies of bone marrow mononuclear cells
Pharmacokinetics (PK) effects of TCP in plasma when combined with ATRA | Baseline, Cycle 1, Cycle 2, 30 Days (+/-10 days) Post-End of Treatment
  Pharmacokinetics (PK) parameters will be determined using serial blood sampling at specified time points to determine PK effects of TCP in plasma when combined with ATRA. Non-compartmental methods of analysis will be used to determine TCP PK parameters following oral dosing of patients in Cycle 1. The following will be calculated: Observed maximum concentration (Cmax), the time at which Cmax occurred (Tmax), the area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC24hr), the terminal disposition phase half-life (t1/2).
Pharmacodynamic (PD) effects of TCP in peripheral blood and bone marrow when combined with ATRA. | Baseline, Cycle 1, Cycle 2, 30 Days (+/-10 days) Post-End of Treatment
  Pharmacodynamics (PD) measurements will be obtained from serial blood and bone marrow sampling at specified time points to describe the PD effects of TCP when combined with ATRA. The following will be measured: Expression of CD11b by flow cytometry, gene expression analysis of leukemic blasts, measurement of Retinoic acid receptor alpha (RARα) and lysine (K)-specific demethylase 1A (LSD1) within leukemic blasts, leukemic engraftment of treated cells in immunodeficient mice.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Watts, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tayari MM, Santos HGD, Kwon D, Bradley TJ, Thomassen A, Chen C, Dinh Y, Perez A, Zelent A, Morey L, Cimmino L, Shiekhattar R, Swords RT, Watts JM. Clinical Responsiveness to All-trans Retinoic Acid Is Potentiated by LSD1 Inhibition and Associated with a Quiescent Transcriptome in Myeloid Malignancies. Clin Cancer Res. 2021 Apr 1;27(7):1893-1903. doi: 10.1158/1078-0432.CCR-20-4054. Epub 2021 Jan 25. PMID 33495312